CLINICAL TRIAL: NCT01781234
Title: Efficacy Study of Intranasal Insulin to Treat Tobacco Abstinence Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ajna Hamidovic (Other)
Responsible Party: Sponsor-Investigator, Ajna Hamidovic, Assistant Professor, University of New Mexico
Organization: University of New Mexico (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNM-246
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Tobacco Abstinence Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Insulin (Experimental): Intranasal Insulin
  Interventions: Drug: Intranasal Insulin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Insulin
  Arms: Intranasal Insulin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate safety and efficacy of intranasal insulin in abstinent smokers. Groups' (placebo vs. insulin) cognitive function and stress response will be compared.

ELIGIBILITY:
Inclusion Criteria:

* smokers (>10 cig/day) for the past 1 year
* normosmic olfactory function

Exclusion Criteria:

* previous/current use of insulin
* current Diagnostic and Statistical Manual-IV-Revised (DSM-IV-R) Axis I disorder
* current pregnancy (or lactation)
* lifetime history of endocrine disease
* excessive alcohol use (>25 standard units of alcohol/week)
* current use of illicit drugs
* current use of a smoking cessation aid (NRT, Chantix or Wellbutrin), or a psychotropic agent
* local infections, inflammation, structural abnormalities, or other nasal pathology
* current use of any medications administered intranasally, including intranasal steroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UNM College of Pharmacy, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Insulin: Group receiving active treatment
- Placebo: Group receiving placebo
Period: Overall Study
Arm/Group | Intranasal Insulin | Placebo
Started | 27 | 24
Completed | 18 | 21
Not Completed | 9 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Insulin | Placebo | Total
Number analyzed (Participants) | 16 | 21 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 21 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.75 (13.23) | 40.19 (13.74) | 37.34694 (12.45417)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 10
  Not Hispanic or Latino | 14 | 13 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 6 | 15
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 6 | 13 | 19
Region of Enrollment [Number; unit: participants]
  United States | 16 | 21 | 37

OUTCOME MEASURES:

1. Primary Outcome: Episodic Memory
Description: California Verbal Learning Task Number of Words Learned Higher Values Mean Better Outcome
Time Frame: 90 minutes
Measure: Mean (Standard Error); unit: number of words recalled
Arm/Group | Intranasal Insulin | Placebo
Number analyzed (Participants) | 16 | 21
number of words recalled | 11.6 (0.3) | 10.0 (0.3)

2. Primary Outcome: Salivary Cortisol
Time Frame: 90 minutes
Measure: Mean (Standard Error); unit: mcg/dL
Arm/Group | Intranasal Insulin | Placebo
Number analyzed (Participants) | 16 | 21
mcg/dL | 0.23 (0.02) | 0.13 (0.01)

3. Other Pre Specified Outcome: Nicotine Craving (Measured by Questionnaire of Smoking Urges)
Description: Questionnaire of Smoking Urges; Total Range= 10-70; Higher values represent worse outcome
Time Frame: 90 minutes
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intranasal Insulin | Placebo
Number analyzed (Participants) | 16 | 21
units on a scale | 30.48 (1.42) | 43.44 (1.39)

ADVERSE EVENTS:
Arm/Group | Intranasal Insulin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24
Other Adverse Events (participants affected / at risk) | 25/27 | 13/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Insulin (N=27) | Placebo (N=24)
Rhinorrhea (General disorders) | 2 (2) | 1 (1) — Nasal Occurrences
Smell (General disorders) | 8 (10) | 1 (1) — Nasal Occurrences
Tingling (General disorders) | 4 (5) | 0 (0) — Nasal Occurrences
Irritation (General disorders) | 7 (9) | 0 (0) — Nasal Occurrences
Sneezing (General disorders) | 2 (2) | 0 (0) — Nasal Occurrences
Numbness (General disorders) | 3 (5) | 0 (0) — Nasal Occurrences
Burning (General disorders) | 2 (2) | 1 (1) — Nasal Occurrences
Sensitivity (General disorders) | 1 (2) | 0 (0) — Nasal Occurrences
Pressure (General disorders) | 0 (0) | 1 (1) — Nasal Occurrences
Congestion (General disorders) | 1 (1) | 0 (0) — Nasal Occurrences
Bleeding (General disorders) | 1 (1) | 0 (0) — Nasal Occurrences
Dryness (General disorders) | 1 (1) | 0 (0) — Nasal Occurrences
Pressure (ears) (General disorders) | 0 (0) | 1 (1) — Other Occurrences
Pressure (eye) (General disorders) | 0 (0) | 1 (1) — Other Occurrences
Dizziness (General disorders) | 6 (7) | 0 (0) — Other Occurrences
Taste (General disorders) | 0 (0) | 1 (1) — Other Occurrences
Sweating (General disorders) | 4 (4) | 1 (1) — Other Occurrences
Bruising (General disorders) | 0 (0) | 1 (2) — Other Occurrences
Headache (General disorders) | 2 (2) | 0 (0) — Other Occurrences
Stomach Pain (General disorders) | 1 (1) | 0 (0) — Other Occurrences
Blurry Vision (General disorders) | 0 (0) | 1 (1) — Other Occurrences
Tingling (throat) (General disorders) | 0 (0) | 1 (1) — Other Occurrences
Confusion (General disorders) | 7 (7) | 2 (2) — Other Occurrences
Numbness (arm) (General disorders) | 1 (1) | 1 (1) — Other Occurrences
Tingling (mouth) (General disorders) | 0 (0) | 3 (3) — Other Occurrences
Cold (General disorders) | 0 (0) | 1 (1) — Other Occurrences
Shaking (General disorders) | 2 (2) | 1 (1) — Other Occurrences
Anxiety (General disorders) | 0 (0) | 1 (1) — Other Occurrences
Itchiness (General disorders) | 1 (1) | 0 (0) — Other Occurrences
Diarrhea (General disorders) | 1 (1) | 0 (0) — Other Occurrences
Difficulty Breathing (General disorders) | 1 (1) | 1 (1) — Other Occurrences
Fatigue (General disorders) | 0 (0) | 1 (1) — Other Occurrences

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes